CLINICAL TRIAL: NCT01888107
Title: Maintenance of Clinical Response With Risperidone Long Acting Injectable (R-LAI) in Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Maintenance of Efficacy With Risperidone Long Acting Injectable (R-LAI) in Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004993; 2004-000830-35 (EudraCT Number)
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Antipsychotics; Risperidone; Long-acting injectable
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risperidone Long-acting Injectable (LAI) (Experimental): Risperidone LAI will be administered in dosages of 25, 37.5, and 50 mg.
  Interventions: Drug: Risperidone Long-acting Injectable (LAI) 25 mg; Drug: Risperidone LAI 37.5 mg; Drug: Risperidone LAI 50 mg

INTERVENTIONS:
Drug: Risperidone Long-acting Injectable (LAI) 25 mg — Risperidone LAI will be administered as a gluteal intramuscular injection given every 2 weeks for 52 weeks.
Drug: Risperidone LAI 37.5 mg — Risperidone LAI will be administered as a gluteal intramuscular injection given every 2 weeks for 52 weeks.
Drug: Risperidone LAI 50 mg — Risperidone LAI will be administered as a gluteal intramuscular injection given every 2 weeks for 52 weeks.

SUMMARY:
The purpose of this study is to assess the maintenance of antipsychotic efficacy and safety of risperidone long-acting injectable (RLAI) in patients with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) or schizoaffective (a mixed psychiatric disorder relating to a complex psychotic state that has features of both schizophrenia and a mood disorder such as bipolar disorder) disorder who were receiving treatment with any antipsychotic medication and who required a long-term antipsychotic therapy. The secondary aim is to investigate prospectively (a study that starts with the present condition of a population of individuals and follows them into the future) the prevalence of patients who met standardized remission criteria (according to Andreasen et al. criteria) and the psychopathological, psychosocial and subjective predictors of achieving remission.

DETAILED DESCRIPTION:
This is a prospective, open-label, (all people know the identity of the intervention), single-arm study conducted at 47 sites in Italy between January 2005 and April 2007. Approximately 338 patients with schizophrenia or schizoaffective disorder who were receiving treatment with any antipsychotic medication and who required a long-term antipsychotic therapy will be switched directly to RLAI without an oral risperidone run-in (the elapsed time before a trial is started when no treatment is given to patients in the study). They will be considered either not optimally treated or symptom-free. Patients will be either not hospitalized or living in residential structures at the time of the enrollment as well as throughout the study. The maximum duration of study participation will be 52 weeks. Patient safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Required long-term antipsychotic therapy at the time of recruitment
* Symptomatically stable and taking the same dose of antipsychotic agents for at least one month before the baseline visit (considered stable if there have been no appreciable change in symptoms over the previous month, regardless of the severity of their symptoms)
* Patients or their legal representatives provided their written informed consent prior to enrollment in the study

Exclusion Criteria:

* Patients who had received clozapine during the previous 3 months
* Participated in an investigational drug trial in the previous 30 days
* Previously been shown to be either intolerant or non-responsive to risperidone therapy
* Presence of a serious unstable medical condition, such as a history or current symptoms of tardive dyskinesia or a history of neuroleptic malignant syndrome
* Pregnant or breast-feeding; female patients of childbearing potential not using adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2005-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) total and subscales score | Baseline and after 4, 12, 26, 38 and 52 weeks
  Maintenance= Symptom severity assessed with PANSS scale vs baseline (Total, positive, negative, general psychopathology and cognitive cluster score); Remission= percentage of patients with 8 specific items PANSS simultaneously scoring <= 3 for at least 6 months

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) scale | Baseline
  This measure is used to evaluate disease severity at baseline (Visit 1).
Change from Baseline in Clinical Global Impression-Change (CGI-C) scale | Baseline and after 4, 12, 26, 38 and 52 weeks
  This measure is used to evaluate disease severity at the other time points (Visits 2 to 6).
Change from Baseline in Global Assessment of Functioning (GAF) | Baseline and after 4, 12, 26, 38 and 52 weeks
  GAF is a 100-point tool rating overall psychological, social and occupational functioning of adults. The higher score range (91-100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (1-10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death. Lower scores indicate worsening.
Change from Baseline in Drug Attitude Inventory (DAI 30) | Baseline and after 4, 12, 26, 38 and 52 weeks
  Personal attitude towards risperidone long-acting injectable treatment is rated by a subjective questionnaire that is administered at each study visit (1 through 6).
The number of patients who experience adverse events as a measure of safety and tolerability. | Baseline and after 4, 12, 26, 38 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.

REFERENCES:
- See also: Maintenance of clinical response with risperidone long-acting injectable (R-LAI) in subjects with schizophrenia or schizoaffective disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1372&filename=CR004993_CSR.pdf